CLINICAL TRIAL: NCT07293988
Title: Clinical, Biomechanical, Histo-immunological and Radiological Characterization of the Effects of Two Gastrocnemius Stretching Programs in Adult Patients With Spastic Paresis Following Cerebral Palsy: MYOSPAS-CP, a Randomized Controlled Study
Brief Title: Spastic Myopathy in Adults With Cerebral Palsy
Acronym: MYOSPAS-IMC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuroloco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-A00041-38; 2019-004945-33 (EudraCT Number)
Record Dates: First submitted 2025-11-26; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy (CP)
Keywords: cerebral palsy; fascicle length; spastic myopathy; micro-invasive biopsy; daily self-stretch posture; muscle volume; muscle thickness; fiber diameter; fiber type; myosin isoform chain; MRI; elastography; stiffness; shear modulus; spastic cocontraction; paresis; gait speed; micro-tester; gastrocnemius
MeSH Terms: conditions — Cerebral Palsy; Paresis

STUDY DESIGN:
Intervention Model Description: In the interventional group, subjects will follow a Guided Self-rehabilitation program based on daily high-load gastrocnemius self-stretching postures (10 minutes/day) and phasic maximal dorsiflexion efforts In the control group, subjects follow their rehabilitation sessions (conventional therapy) as before their enrollment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Self-rehab group (Experimental): In the interventional group, subjects will follow a Guided Self-rehabilitation program based on daily high-load gastrocnemius self-stretching postures (10 minutes/day) and phasic maximal dorsiflexion efforts
  Interventions: Behavioral: Guided Self-rehabilitation Contract
- Control group (Other): In the control group, subjects follow their rehabilitation sessions (conventional therapy) as before their enrollment
  Interventions: Behavioral: Conventional therapy group

INTERVENTIONS:
Behavioral: Guided Self-rehabilitation Contract — Participants randomized to the intervention arm will receive a one-year individualized program based on the Guided Self-Rehabilitation Contract (GSC) method. A physiotherapist specifically trained in GSC will supervise all 20 patients. The therapist will conduct monthly 1.5-hour home visits, supplemented as needed by intermediate webcam or telephone consultations.
  The GSC method aims to increase the patient's knowledge, responsibility, and active involvement in their rehabilitation. Its core psychological mechanism is the use of a daily quantified logbook (paper, electronic, or the i-GSC™ smartphone/tablet application). Patients must record daily stretching time per muscle and the number of active movements performed in each series. The therapist explains that maintaining this logbook is a central component of the therapeutic contract. At each visit, the logbook is reviewed to enhance data accuracy, monitor motivation, reinforce adherence, and provide positive feedback-mechanisms show
  Arms: Guided Self-rehab group
Behavioral: Conventional therapy group — In this group, subjects follow their rehabilitation sessions as before their enrollment. Conventional physiotherapy will typically consist of one to three sessions per week, delivered either in a private outpatient practice or at the patient's home, depending on the medical prescription. Session duration and therapeutic content may vary, reflecting routine real-life practice. Quantitative and qualitative data regarding conventional physiotherapy will be collected for all subjects throughout the study
  Arms: Control group

SUMMARY:
Cerebral palsy (CP) is indeed the result of a central neurological lesion, but it also involves a lesser-known muscular condition that we refer to as spastic myopathy. This condition is likely the consequence of relative immobilization and underuse of the muscles in the affected limbs and, through a vicious cycle, it in turn plays a major role in movement difficulties. Among the muscles involved are the plantar flexors, whose extensibility decreases from the earliest years of the child's life.

The BIOTN research team (UR7377; Université Paris-Est Créteil; Dr M. Pradines, Prof. J.-M. Gracies, CHU Henri Mondor, Créteil), supported by the Fondation pour la Paralysie Cérébrale, is conducting a randomized controlled study aimed, on the one hand, at characterizing in these individuals the genetic, histological, radiological, mechanical, physiological, and clinical changes in the calf muscle, and on the other hand, at exploring the reversibility of these alterations by comparing the effects of two types of rehabilitation after one year.

This study will provide essential insights for the development of specific and adapted rehabilitation strategies designed to improve the living conditions of individuals with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy (CP), resulting from a perinatal central neurological lesion, leads not only to lifelong motor impairment but also to a specific muscular disorder: spastic myopathy. This condition is characterized by early and progressive structural changes including decreased passive extensibility (XV1), reduced muscle fiber diameter, decreased number of sarcomeres in series, and hypertrophy of the endomysium and perimysium. In children, impaired gastrocnemius growth-quantified by reduced medial gastrocnemius muscle volume-appears before age 3 and precedes both hyperactivity and fixed stiffness. However, the long-term consequences of decades of underuse on the mechanical, histological, and morphometric properties of the gastrocnemius in adults with IP remain insufficiently explored.

Stretching, although widely prescribed, lacks standardized parameters, and its long-term effectiveness in adults with IP has never been formally evaluated. Evidence suggests that muscular plasticity requires high-load stretching and ≥10 minutes per muscle per day. Preliminary studies using Guided Self-Rehabilitation Contracts (GSCs) demonstrated significant gains in extensibility and function, while a randomized controlled trial in adults with acquired hemiparesis showed increased fascicle length, increased muscle thickness, and improved gait speed after one year of high-load self-stretching, supporting the reversibility of molecular pathways driving contracture.

This single-blind randomized controlled trial includes 40 adults with IP, randomized to: (1) conventional physiotherapy alone, or (2) conventional physiotherapy + a one-year daily GSC-based high-load gastrocnemius self-stretching program (10 minutes/day + phasic maximal dorsiflexion efforts). Multi-scale assessments span six analytical domains: clinical measures (XV1, XV3, XA; gait speed; SF-36), in vivo tissue biomechanics (resistance torque, passive energy, fascicle length, muscle thickness), functional and neurophysiological biomechanics (agonist-antagonist recruitment during gait), MRI morphometry (volume, intramuscular fat, edema), in vitro biomechanics (compressibility, strain, rupture stress), and genetic/histological markers (satellite cells, expression profile of 57 myogenic genes). Micro-invasive biopsies of both limbs will be performed at J1 and M12.

The primary outcome is maximal barefoot 10-meter gait speed. Secondary outcomes will characterize, chronologically and mechanistically, the trajectory of spastic myopathy and the potential of long-term high-load stretching to partially reverse its pathogenic processes.

ELIGIBILITY:
Inclusion Criteria:

* Hemiparesis or diparesis resulting from a cerebral lesion occurring during the perinatal period (cerebral palsy).
* Gastrocnemius extensibility XV1 < 100° (XV1, Tardieu Scale).
* Maximum barefoot walking speed (AT10) between 0.3 and 1.2 m/s.
* Written informed consent to participate in the study.

Exclusion Criteria:

* Botulinum toxin injections in the medial gastrocnemius within less than 3 months prior to study inclusion.
* Cognitive impairment preventing participation in the GSC program or in the study.
* Patients under legal guardianship or conservatorship.
* Known hemostasis disorders.
* Hypersensitivity to allergens.
* Presence of a metallic intraocular foreign body (accidental fragments or others), a pacemaker, a neurostimulator (pain treatment), a cochlear implant, or, more generally, any implanted electronic medical device that cannot be removed; presence of a metallic cardiac valve in the study participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Maximal ambulation speed over 10 meters | Day 1, Month 6, Month 12
  Maximal ambulation speed over 10 meters, barefoot

SECONDARY OUTCOMES:
Plantar flexor clinical extensibility (XV1) | Day 1, Month 6, Month 12
  Passive ankle dorsiflexion were assessed using standardized Tardieu Scale procedures. XV1 was measured during a very slow, strong passive stretch of the gastrocnemius with the patient supine, knee extended. The stretch was performed over 3-5 seconds to minimize stretch-reflex activation, and the maximal angle at which soft-tissue resistance could no longer be overcome was recorded as the passive maximal dorsiflexion range (XV1).
Plantarflexor spasticity | Day 1, Month 6, Month 12
  XV3 was obtained under identical positioning as XV1 but during a rapid stretch (V3). To ensure the muscle was fully relaxed prior to the fast movement, the examiner performed several quick oscillatory pre-movements in the opposite direction. The angle of catch or clonus during the fast stretch defined XV3.
Active dorsiflexion (XA) | Day 1, Month 6, Month 12
  XA represented maximal active dorsiflexion, measured with the patient supine and knee extended, reflecting both passive and active constraints imposed by the gastrocnemius.
LG Young modulus | Day 1, Month 6, Month 12
  Participants were assessed using a share wave elastography system while seated in an isokinetic ergometer (trunk at 60°, knee extended, ankle fixed). The lateral gastrocnemius (GL) shear modulus (µGL) were measured through nine sites (superior, middle, inferior, medial, medium, lateral). Measurements were performed under two ankle positions: 40° plantarflexion (non-stretched LG) and 80% of individual XV1-GAS (stretched LG). For each site and condition, 10-second cine loops were recorded (a validated acquisition method), yielding 10 videos per participant. Each video was then divided into 10 DICOM frames to obtain reliable µGL estimates. Image processing and µGL extraction were performed using MATLAB®.
LG fascicle length | Day 1, Month 6, Month 12
  Participants were assessed using a high frequency ultrasound system while seated in an isokinetic ergometer (trunk at 60°, knee extended, ankle fixed). Structural ultrasound images at the middle/medium location were analyzed to derive fascicle length
LG Tickness | Day 1, Month 6, Month 12
  Participants were assessed using a hifh frequency ultrasound system while seated in an isokinetic ergometer (trunk at 60°, knee extended, ankle fixed). Structural ultrasound images at the middle/medium location were analyzed to determine muscle thickness
LG Muscle volume | Day 1, Month 12
  A high-field 3T MRI examination of both the paretic and contralateral lateral gastrocnemius muscles will be performed using a flexible surface coil positioned around the patient's calves. Muscle volume will be quantified from a series of continuous axial T1-weighted slices acquired along the full length of the calf.
Intramuscular fat percentage | Day 1, Month 12
  A high-field 3T MRI examination of both the paretic and contralateral lateral gastrocnemius muscles will be performed using a flexible surface coil positioned around the patient's calves. Intramuscular fat percentage will be estimated using a Dixon sequence, allowing reliable separation of water and fat signals.
LG hyperelastic behavior under compression | Day 1, Month 12
  A micro-invasive muscle biopsy using a Weil-Blakesley forceps will be performed twice, one year apart, on both the paretic and contralateral lateral gastrocnemius of each participant. This technique will be carried out by a trained investigator under local anesthesia. The biopsy will target the LG muscle belly, yielding approximately 30 mg of tissue for in vitro biomechanical analysis. Using an MTS Insight machine, fresh muscle fragments will undergo sequential uniaxial tensile and compressive relaxation tests. These procedures will enable detailed quantification of hyperelastic behavior under compression.
LG fiber-type composition | Day 1, Month 12
  From biopsies, ~30 mg of tissue will be cryosectioned to visualize 400-500 fibers. Immunohistochemistry will determine fiber-type composition (fast/slow myosin)
LG endo-/perimysial fibrosis | Day 1, Month 12
  From biopsies, ~30 mg of LG tissue will be cryosectioned to visualize 400-500 fibers. Standard stainings (H&E, Gomori Trichrome, COX, Sirius Red) will assess endo-/perimysial fibrosis.
LG genetic expression | Day 1, Month 12
  From biopsies, ~30 mg of LG tissue will be used to examine the expression of 57 genes related to skeletal muscle structure, myogenic differentiation, metabolic regulation, and atrophy pathways. RNA will be extracted with the Nano PreAMP kit (Qiagen), and gene expression profiled using the RT² Profiler™ PCR Array - Human Skeletal Muscle Development & Disease. The targeted gene groups include markers of the dystrophin-glycoprotein and titin complexes, fast and slow fiber signatures, energy metabolism, myogenesis (MYOD1, MYOG, PAX3/7), atrophy/autophagy (FBXO32, TRIM63, TNF)
LG spastic cocontraction | Day 1, Month 12
  Participants will be equipped with bilateral surface EMG electrodes on the tibialis anterior and lateral gastrocnemius (ME6000, 16-channel WiFi system; 1000 Hz). LG spastic cocontraction will be quantified during maximal dorsiflexion effort. When technically feasible, Mmax will be used as an alternative denominator of MVC in these ratios through tibial nerve stimulation
Plantar/dorsiflexion strength | Day 1, Month 6, Month 12
  Participants will be positioned in the ConTrex device, at two ankle positions (40° plantarflexion = relaxed GL; and 80% XV1-GAS = stretched GL). The maximal strength in dorsiflexion and plantarflexion will be quantified by the isokinetic ergometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Maud Pradines, Créteil, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided